CLINICAL TRIAL: NCT01466803
Title: Effects of Voriconazole on the Pharmacokinetics and Pharmacodynamics of Oral Buprenorphine: A Two-phase Cross-over Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Mari Fihlman, MD, Turku University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Oralbupre
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Buprenorphine; Vorikonazole; Interactions; Pharmacokinetics; Pharmacodynamics; Voriconazole

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Vorikonazole (Active Comparator): The subject will be given vorikonazole twice a day for 5 days prior to the study. The dose will be 400 mg twice a day on day one ans 200 mg twice a day on days 2-5.
  Interventions: Drug: Vorikonazole
- Placebo (Placebo Comparator): The subjects will be given placebo twice a day for 5 days prior to the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — The subjects will be given placebo twice a day for 5 days prior to the study
  Arms: Placebo
Drug: Vorikonazole — The subject will be given vorikonazole twice a day for 5 days prior to the study. The dose will be 400 mg twice a day on day one ans 200 mg twice a day on days 2-5.
  Arms: Vorikonazole

SUMMARY:
Variability in drug response can be due to either pharmacokinetic or pharmacodynamic factors. The reasons why people differ in pharmacokinetics or pharmacodynamics are manifold and include, e.g., genetic factors, diseases, age and concomitantly administered drugs. Oxidation reactions are dominant in the metabolism of drugs and cytochrome P-450 enzymes (CYP) have been recognized as chief contributors (Guengerich 1992). We have previously shown that drug interactions mediated by the inhibition of CYP enzymes may be of major clinical significance (Olkkola et al. 1993; Olkkola et al. 1994; Varhe et al. 1994; Olkkola et al. 1999; Palkama et al. 1999; Jokinen et al. 2000).

Buprenorphine undergoes extensive first-pass metabolism and has low oral bioavailability of 15 % (Cone et al. 1984). Bioavailability following sublingual administration of buprenorphine is higher, 50-60 % (Nath et al. 1999). After high sublingual doses of buprenorphine (8-24 mg), peak plasma concentrations are reached in 1 hour (McAleer et al. 2003, Ciraulo et al. 2006) and after low sublingual doses (0.4 mg) they are reached in approximately 3 h (Billingham 1981). Approximately two-thirds of a buprenorphine dose is excreted unchanged, and the rest is metabolized in the liver and intestinal wall. N-dealkylation of buprenorphine mainly via CYP3A but also CYP2C8 yields norbuprenorphine, and glucuronidation yields buprenorphine-3-glucuronide (Cone et al. 984). Norbuprenorphine is excreted in the urine after subsequent conjugation. 80-90 % of buprenorphine is excreted by the biliary system and enterohepatic circulation (Brewster et al. 1984)

Although few interaction studies of high-dose buprenorphine and antiretrovirals have been conducted (McCance-Katz EF et al. 2007), the effect of CYP3A inhibitors on the pharmacokinetics of low-dose buprenorphine is unknown. Because the use of buprenorphine in pain management is increasing after the introduction of transdermal buprenorphin patches to the market, it is clinically relevant to study and quantify possible interactions of buprenorphine with inhibitors of its CYP3A-mediated metabolism such as voriconazole.

This study is aimed to examine the possible interactions of oral buprenorphine with voriconazole.

Twelve male or female adult non-smoking subjects aged 18-40 years with body weights within ±15% of the ideal weight for height will be recruited for the study. The subjects will be submitted to physical examination, determination of previous or present chronic diseases, and comprehensive laboratory testing to ascertain that they are in good health. The subjects will fill in a modified Finnish version of the Abuse Questions (Michna et al. 2004) to assess their vulnerability for opioid abuse. Laboratory screening will include CBC (including hemoglobin, hematocrit, differential WBC, platelet count), SGOT, SGPT, alkaline phosphatase, BUN and creatinine, and for women a pregnancy test. Urine will be screened for glucose, proteins and drugs with addiction potential. Blood pressure in sitting position must be within normal limits. Base line ECG must be normal.

Placebo and voriconazole should always be ingested with food, except the first dose on day 5.

On day 5, the challenge dose of 0.2 or 3.6. mg of oral buprenorphine (Temgesic, Schering-Plough) will be administered at 11.00, i.e. 1 h after the last dose of placebo or voriconazole. The dose is 3.6 mg after placebo and 0.2 mg after voriconazole. If necessary, naloxone (Naloxone B. Braun, Braun) will be given in sufficient doses to counteract the severe adverse effects of buprenorphine. For nausea and vomiting, intravenous tropisetron will used, if needed.

The volunteers will fast at least 8 h before the administration of buprenorphine and they will have a standard meal 4 h and 8 h afterwards. Ingestion of alcohol, coffee, tea, cola, energydrinks and grapefruit juice is not allowed during the test days, nor is smoking permitted.

The interval between the study phases will be four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-40
* Body weight within ±15% of the ideal weight for height

Exclusion Criteria:

* A previous history of intolerance to the study drugs or to related compounds and additives
* Concomitant drug therapy of any kind for at least 14 days prior to the study
* Existing or recent significant disease
* History of hematological, endocrine, metabolic or gastrointestinal disease, including gut motility disorders
* History of asthma or any kind of drug allergy
* Previous or present alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements
* A positive test result for urine toxicology
* A "yes" answer to any one of the Abuse Questions
* Pregnancy or nursing
* Donation of blood for 4 weeks prior and during the study
* Special diet or life style conditions which would compromise the conditions of the study or interpretation of the results
* Participation in any other studies involving investigational or marketed drug products concomitantly or within one month prior to the entry into this study
* Smoking for one month before the start of the study and during the whole study period
* Any history of coagulation abnormality, also in first degree relatives

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Concentration of buprenorphine and its metabolites in plasma and urine Concentration of buprenorphine and its metabolites in plasma and urine | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 and 20 hours after administration of buprenorphine

SECONDARY OUTCOMES:
Pharmacodynamic effects | 1, 2,3, 4, 5, 6, 8, 10, 12, hours after administration of buprenorphine
  The psychomotor effects on buprenorphine will be assessed with the measurement of pupil size, Maddox wing test and digit symbol substitution test
Analgesia | 1, 2, 3, 4, 5, 6, 8, 10, 12 hours after the administration of buprenorphine
  The analgesic effect of buprenorphine will be evaluated using the cold pressor test. Briefly, the subject's hand is immersed into ice-cold water of + 4° C up to the wrist. The subject is told to keep his or her hand in the water and to report when the cold sensation becomes painful. Cold pain threshold is defined as the latency from the immersion of the hand to the subject's first report of pain. Cold pain intensity is assessed at 30 s intervals following immersion of the hand in cold water for up to 60s . A verbal numerical rating scale of 0-100 will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland